CLINICAL TRIAL: NCT03738891
Title: A Feasibility Study to Evaluate Electromagnetic Muscle Stimulation and CoolSculpting for Abdominal Contouring
Brief Title: CoolSculpting and EMS for the Abdomen
Acronym: ECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA18-003
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Electromagnetic Muscle Stimulation (EMS) only - Cohort 1 (Experimental): Subjects in this group will be treated with 4 sessions of EMS. CoolSculpting will not be used.
  Interventions: Device: Electromagnetic Muscle Stimulation alone
- Electromagnetic Muscle Stimulation (EMS) followed by CoolSculpting- Cohort 2 (Experimental): Following 4 sessions of EMS, subjects will receive 3-6 cycles of CoolSculpting.
  Interventions: Device: EMS followed by CoolSculping
- CoolSculpting only - Cohort 3 (Experimental): Subjects in this arm will receive 3-6 cycles of CoolSculpting treatments.
  Interventions: Device: Zeltiq CoolSculpting System alone
- CoolSculpting followed by Electromagnetic Muscle Stimulation (EMS )- Cohort 4 (Experimental): Subjects in this group will have 3-6 cycles of CoolSculpting followed by 4 EMS sessions.
  Interventions: Device: CoolSculpting followed by EMS

INTERVENTIONS:
Device: Zeltiq CoolSculpting System alone — The CoolSculpting System will be used to perform the treatments in Cohort 3.
  Other Names: CoolSculpting
  Arms: CoolSculpting only - Cohort 3
Device: Electromagnetic Muscle Stimulation alone — The EMS device(s) alone are used in Cohort 1.
  Other Names: EMS
  Arms: Electromagnetic Muscle Stimulation (EMS) only - Cohort 1
Device: EMS followed by CoolSculping — Cohort 2 group will be treated with EMS followed by CoolSculpting
  Arms: Electromagnetic Muscle Stimulation (EMS) followed by CoolSculpting- Cohort 2
Device: CoolSculpting followed by EMS — Cohort 4 will be treated first with CoolSculpting, followed by EMS.
  Arms: CoolSculpting followed by Electromagnetic Muscle Stimulation (EMS )- Cohort 4

SUMMARY:
Evaluate the use of Electromagnetic Muscle Stimulation as an adjunctive treatment to CoolSculpting.

ELIGIBILITY:
Inclusion Criteria

* Male and female subjects > 22 years of age and ≤65 years of age.
* Subject has not had weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject agrees to refrain from any new abdominal training exercises during the course of the study.
* BMI ≤ 30 kg/m^2 as determined at screening.
* Abdominal skin fold thickness 2.0 to 5.0 cm, as measured by caliper below umbilicus.
* Cohort 4 only: Subject participated in protocol ZA18-003 in Cohort 3, and received the CoolSculpting treatment no more than 6 months prior.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction, body contouring and/or skin tightening procedure in the area of intended treatment within the past 12 months.
* Subject has numbness, tingling or other altered sensation in the treatment area.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has not had an intrauterine contraceptive device inserted or removed within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the Investigator's opinion may increase the subject's risk of bruising.
* Subject has known sensitivity or allergy to isopropyl alcohol and propylene glycol, or latex.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites, that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has a metal implant or active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Subject has been involved in any type of abdominal muscle training program within the previous 6 months.
* Subject has pulmonary insufficiency.
* Subject has a cardiac disorder.
* Subject has a malignant tumor.
* Subject has been diagnosed with epilepsy.
* Subject currently has a fever.
* Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, NP, Study Director — Zeltiq Aesthetics
Locations (4):
- United States (4):
  - Marina Plastic Surgery, Marina del Rey, California
  - Innovation Research Center, Pleasanton, California
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Aesthetic Solutions, P.A., Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kilmer SL, Cox SE, Zelickson BD, Bachelor EP, Gamio S, Ostrowski R, Pham LD, Stevens WG. Feasibility Study of Electromagnetic Muscle Stimulation and Cryolipolysis for Abdominal Contouring. Dermatol Surg. 2020 Oct;46 Suppl 1(1):S14-S21. doi: 10.1097/DSS.0000000000002420. PMID 32976168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 50 participants enrolled into Cohorts 1, 2, and 3. One subject enrolled in Cohort 3, received the treatment and completed all follow-up visits per Cohort 3 before subsequently rolling over to, and receiving treatment planned for Cohort 4. No other subjects were enrolled in Cohort 4. Efficacy data for Cohort 4 was excluded from analysis to avoid the perception of enhancing study enrollment. Data from this participant's treatment in Cohort 3 was included in all endpoint analyses.
Groups:
- Cohort 1-EMS Only: Participants in this group were treated with 4 sessions of Electromagnetic Muscle Stimulation (EMS). CoolSculpting was not used.
- Cohort 2 - EMS Followed by CoolSculpting: Participants were treated with EMS (4 sessions) followed by 1 CoolSculpting treatment (3-6 cooling cycles)
- Cohort 3 - CoolSculpting Only: Participants were treated with 1 CoolSculpting treatment (3-6 cooling cycles)
- Cohort 4: Participants were treated with 1 CoolSculpting treatment (3-6 cooling cycles) followed by 4 sessions of EMS.
Period: Initial Cohort Assignment
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only | Cohort 4
Started | 20 | 20 | 10 | 0
Completed | 20 | 20 | 10 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Subsequent Cohort Assignment
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only | Cohort 4
Started | 0 | 0 | 0 | 1 (One subject was enrolled in Cohort 3, received CoolSculpting treatment, and completed all follow-up visits for that cohort before subsequently rolling over to, and receiving EMS treatment per Cohort 4, permitted by an amendment to the protocol. No other subjects were enrolled in Cohort 4.)
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data gathered and presented here by all participants enrolled with evaluable data. One subject enrolled in Cohort 3, received the treatment and completed all follow-up visits per Cohort 3 before subsequently rolling over to, and receiving treatment planned for Cohort 4. No other subjects were enrolled in Cohort 4. Baseline characteristics presented here are for all subjects at the time they were initially enrolled in the study.
Groups:
- Cohort 2 - EMS Followed by CoolSculpting: articipants were treated with EMS (4 sessions) followed by 1 CoolSculpting treatment (3-6 cooling cycles)
- Total: Total of all reporting groups
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only | Total
Number analyzed (Participants) | 20 | 20 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.8) | 38.2 (9.3) | 47.7 (7.9) | 42.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 8 | 38
  Male | 4 | 6 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Am. Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Black or African American | 0 | 0 | 0 | 0
  Native Hawaiian or Pac Islander | 0 | 0 | 0 | 0
  Caucasian | 17 | 18 | 8 | 43
  Other | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 10 | 50
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (2.1) | 24.1 (2.3) | 23.9 (2.1) | 23.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Unanticipated Adverse Device Effects (UADE)
Description: The number of UADEs occurring during the study will be tabulated.
Time Frame: Enrollment through the final 12-week follow-up visit.
Population: All Participants who received at least one study treatment. Participants in all cohorts were evaluated for adverse events.
Measure: Number; unit: events
Groups:
- Cohort 2 - EMS and CoolSculpting: Following 4 sessions of EMS, participants received 3-6 cycles of CoolSculpting.
- Cohort 3 - CoolSculpting Only: Participants in this arm received 3-6 cycles of CoolSculpting treatments.
- Cohort 4 - CoolSculpting Followed by EMS: Following 3-6 cycles of CoolSculpting treatments, participants were treated with 4 sessions of EMS.
  Cohort 4 included a single subject who was rolled over after completing Cohort 3 study activities.
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS and CoolSculpting | Cohort 3 - CoolSculpting Only | Cohort 4 - CoolSculpting Followed by EMS
Number analyzed (Participants) | 20 | 20 | 10 | 1
events | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Global Aesthetic Improvement Per Independent Physician Review of Photographs Based on Investigator Global Aesthetic Improvement Scale (GAIS-Independent)
Description: Comparison of pre-treatment- and 12-week post-final treatment photographs by independent physician reviewer. The reviewer was blinded to the method of treatment and study cohort; baseline and 12-week post-treatment photos were not blinded. After Sponsor training, the reviewer entered assessments according to the Global Aesthetic Improvement Scale (GAIS). The GAIS had outcome choices of "very much improved", "much improved", "improved", "no change", "worse", "much worse", or "very much worse", with "very much improved" representing the most aesthetic improvement. Reported here is the sum of participants who were assessed as improved ("Very Much Improved," "Much Improved", and "Improved").
Time Frame: Baseline photos will be compared to images collected at the final 12-week post-treatment follow-up visit.
Population: All enrolled participants in Cohort 1 were included in the efficacy analysis. Cohort 2 excluded 1 participant for weight outside of protocol requirements and 1 subject for lack of 12-week follow-up photos. Cohort 3 excluded 1 participant due to a surgical procedure in the treatment area. Cohort 4 excluded one participant previously enrolled and treated in Cohort 3 (allowed per protocol); participant included in Cohort 3 analysis only.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 - EMS Followed by CoolSculpting: Following 4 sessions of EMS, participants received 3-6 cycles of CoolSculpting.
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only
Number analyzed (Participants) | 20 | 18 | 9
Participants | 16 | 16 | 8

3. Secondary Outcome: Change in Pre-treatment and Post-treatment Abdominal Circumference
Description: Abdominal circumference as measured by 3-Dimensional imaging prior to treatment (baseline) is compared to images collected at the final 12-week post-treatment follow-up visit. Measurements were captured at 3 points including the upper, middle and lower abdomen. All measurements were averaged per subject at the baseline and 12-week visit time points to obtain circumference values. Results for each cohort are shown in millimeters of circumference reduction.
Time Frame: Baseline and final 12-week follow-up visit.
Population: There were no exclusions from efficacy analysis in Cohort 1. One (1) participant in Cohort 2 was excluded from the analysis due to weight outside requirements of the protocol; 1 participant from cohort 3 was excluded due to a surgical treatment; cohort 4 consisted of a single participant treated in cohort 3 and subsequently rolled over to cohort 4 after cohort 3 final follow-up was completed. Cohort 4 was therefore not analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only
Number analyzed (Participants) | 20 | 19 | 9
mm | -4 (16) | -15 (11) | -10 (18)

4. Secondary Outcome: Percentage of Participants With Global Aesthetic Improvement Scale (S-GAIS) Reporting Improvement
Description: Subjects completed a graded 7-point GAIS at 12-week post-final treatment follow-up. The scale consists of the following response options: 3 = Very much improved; 2 = Much improved; 1 = Improved; 0 = No change; -1 = Worse; -2 = Much worse; -3 = Very much worse. Results were tabulated across the three treatment cohorts. Results were calculated in the percentage of the subjects reporting improvement.
Time Frame: Final post-treatment 12-week follow-up visit
Population: All enrolled subjects with a completed S-GAIS at post-treatment 12-week follow-up visit. Cohort 4 was not included in the tabulation as the single subject treated in this cohort had been previously treated in Cohort 3 (allowed per protocol). Results for the single subject treated in both Cohort 3 and Cohort 4 were tabulated with Cohort 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1 - Electromagnetic Muscle Stimulation (EMS) Only: Participants in this group will be treated with 4 sessions of EMS. CoolSculpting will not be used.
- Cohort 2 - Electromagnetic Muscle Stimulation (EMS) Followed by CoolSculpting: Following 4 sessions of EMS, participants will receive 3-6 cycles of CoolSculpting.
- Cohort 3 - CoolSculpting Only: Participants in this arm will receive 3-6 cycles of CoolSculpting treatments.
Arm/Group | Cohort 1 - Electromagnetic Muscle Stimulation (EMS) Only | Cohort 2 - Electromagnetic Muscle Stimulation (EMS) Followed by CoolSculpting | Cohort 3 - CoolSculpting Only
Number analyzed (Participants) | 20 | 19 | 9
percentage of participants | 70 [46 to 88] | 89 [67 to 99] | 100 [66 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time of enrollment through the final 12-week follow-up visit.
Groups:
- Cohort 4 - CoolSculpting Followed by EMS: Following 3-6 cycles of CoolSculpting treatments, participants were treated with 4 sessions of EMS
Arm/Group | Cohort 1-EMS Only | Cohort 2 - EMS Followed by CoolSculpting | Cohort 3 - CoolSculpting Only | Cohort 4 - CoolSculpting Followed by EMS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 0/20 | 2/20 | 1/10 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-EMS Only (N=20) | Cohort 2 - EMS Followed by CoolSculpting (N=20) | Cohort 3 - CoolSculpting Only (N=10) | Cohort 4 - CoolSculpting Followed by EMS (N=1)
Planned hysterectomy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold virus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03738891/Prot_SAP_000.pdf